CLINICAL TRIAL: NCT06974123
Title: A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of Oral Teslanbaicin in Patients With Radiation Proctitis
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.[2024] 37
Record Dates: First submitted 2025-04-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-10

CONDITIONS: Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arm one (Experimental)
  Interventions: Drug: A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of Oral Tesilanbaiju in Patients with Radiation Proctitis; Drug: Teslanbai oral therapy

INTERVENTIONS:
Drug: A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of Oral Tesilanbaiju in Patients with Radiation Proctitis — Patients clinically diagnosed with radiation proctitis of CTCAE grade I-II will receive oral administration. Three dose groups of Teslanbai bacteria are tentatively planned, formulated as capsules with viable bacterial counts per capsule of ≥1107 CFU, 1108 CFU, and 1*109 CFU, respectively. A "3+3" dose-escalation design will be adopted. Each dose group will enroll 3 subjects. If 1 subject experiences a grade ≥3 adverse reaction, 3 additional patients will be added. If 2 subjects exhibit adverse reactions, enrollment into higher dose groups will be discontinued. The final dosage for subsequent use of Teslanbai bacteria will be determined based on efficacy and safety data.
  Approximately 9 subjects are planned for enrollment. After determining the optimal dosage, investigators and sponsors will decide whether to proceed to Phase II based on the study results and external data.
Drug: Teslanbai oral therapy — A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of Oral Tesilanbaiju in Patients with Radiation Proctitis

SUMMARY:
Radiation Proctitis refers to rectal radiation injury caused by radiotherapy for pelvic malignancies. It is classified into Acute Radiation Proctitis (ARP) and Chronic Radiation Proctitis (CRP) based on onset time and disease progression, with a 3-month threshold distinguishing acute from chronic forms. Over 75% of patients undergoing pelvic radiotherapy develop ARP, while 5%-20% progress to CRP. CRP patients experience persistent symptoms and severe late complications such as gastrointestinal bleeding, perforation, obstruction, and fistulas, which pose significant clinical challenges and severely impact quality of life.

Probiotics have long been used in treating radiation proctitis. Radiotherapy disrupts the intestinal microbiome, leading to dysbiosis. Probiotics help restore microbial balance, normalize intestinal pH, and alleviate diarrhea. Commonly used probiotics include Lactobacillus, Bifidobacterium, Enterococcus, and Lactic Acid Bacteria. Clinical studies indicate probiotics significantly reduce radiotherapy-associated diarrhea risk. However, evidence for their efficacy against other symptoms (e.g., hematochezia, anal pain, tenesmus) or severe complications remains limited. A meta-analysis of 904 patients confirmed probiotics outperform placebos in reducing diarrhea incidence and decreasing loperamide use or watery stool frequency during pelvic radiotherapy.

Lactobacillus rhamnosus, a key probiotic in the human gut, colonizes the gastrointestinal tract and improves inflammatory bowel disease (IBD) symptoms by balancing microbiota, enhancing mucosal barriers, modulating immunity, and suppressing inflammation. Studies show it protects mice from radiation-induced intestinal epithelial damage by reducing apoptosis, increasing crypt survival, and shielding epithelial stem cells.

Chronic intestinal inflammation elevates reactive oxygen species (ROS) levels. Excessive ROS oxidizes cellular structures, triggers inflammatory cytokine release, promotes collagen deposition and fibrosis, and accelerates intestinal barrier damage. Reducing ROS may thus aid IBD prevention and treatment. Selenium, a trace element essential for glutathione peroxidase, scavenges ROS. Lactobacillus rhamnosus cultured with nano-selenium enhances selenium bioavailability. Selenium-enriched Lactobacillus rhamnosus may synergistically modulate gut microbiota and lower ROS to suppress inflammation.

Lactobacillus rhamnosus, approved as a food probiotic, has been safely consumed by 2-5 million people daily since the mid-1990s. Teslanbai bacteria, a novel probiotic derived from Lactobacillus rhamnosus (strain CICC 6137 from China Center of Industrial Culture Collection), incorporates nano-selenium via fermentation and freeze-drying. Preclinical studies demonstrate that oral Teslanbai alleviates DSS-induced acute enteritis symptoms, prevents weight loss, improves intestinal ulcers, reduces vascular permeability, and restores barrier function in mice. Treated mice exhibited intact intestinal structures and formed stools. Safety assessments revealed no adverse effects on blood components or major organs, suggesting Teslanbai's potential efficacy against radiation proctitis.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation with signed informed consent form, good compliance, ability to cooperate with diagnosis, treatment, and follow-up; Age ≥18 years (inclusive), regardless of gender; Pathologically confirmed pelvic malignancies (via histology or cytology) requiring pelvic radiotherapy, clinically diagnosed with Grade 1-2 radiation proctitis (per CTCAE criteria); Karnofsky Performance Status (KPS) score ≥60; Expected survival period ≥6 months;

Normal function of major organs, with laboratory values meeting the following criteria:

Absolute neutrophil count (ANC) ≥1.5×10^9/L Platelets ≥75×10^9/L Hemoglobin ≥90g/L Creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) >60 mL/min/1.73m² (Cockcroft-Gault formula) Total bilirubin <1.5×ULN AST/ALT <2.5×ULN (≤5×ULN for subjects with liver metastasis) Albumin (ALB) ≥30g/L INR or prothrombin time (PT) <1.5×ULN (if on anticoagulant therapy, PT must be within the intended therapeutic range).

Exclusion Criteria:

Severe internal and external hemorrhoids; Allergy to any component of the investigational drug; Comorbid inflammatory bowel disease, irritable bowel syndrome, chronic gastrointestinal bleeding, or other diseases potentially associated with chronic diarrhea symptoms; Specific dietary habits prone to causing intestinal symptoms that cannot be modified; Personality or psychiatric disorders, individuals lacking civil capacity or with limited civil capacity; Medical history, conditions, treatments, or laboratory abnormalities that may interfere with trial results or hinder full participation; Other circumstances deemed unsuitable for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of oral administration of Teslancure in patients with radiation proctitis | From enrollment to the end of treatment at 8 weeks
  Efficacy and Safety Follow up
  1. Efficacy Evaluation Plan Frequency : Initial assessment at Day 30 (±3 days) after the first dose, then every 4 weeks (±3 days) thereafter.
     Termination Criteria : Subject death, withdrawal of informed consent, or study completion.
     Assessment Items :
     Physical examination Vital signs (blood pressure, heart rate, temperature, etc.) KPS Score (Karnofsky Performance Status) Patient reported outcomes (EORTC QLQ C30 questionnaire) Concomitant medications/treatments Adverse events (AEs) Laboratory tests (blood tests, biochemistry, etc., as per protocol) Vienna Rectoscopy Score (if applicable)
  2. Safety Follow up Plan (1) Telephone Follow up Time Points : Day 7 (±3 days) and Day 15 (±3 days) after the first dose.
  Content :
  Recording of adverse events (AEs) Assessment of clinical symptom relief

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided